CLINICAL TRIAL: NCT05897567
Title: Effects of Ketogenic Diet on Muscle Hypertrophic Response to Resistance Exercise
Brief Title: Effect of Ketogenic Diet on Muscle Hypertrophy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Padova (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KETO-EX
Record Dates: First submitted 2023-05-18; First posted 2023-06-09 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2023-05

CONDITIONS: Healthy Nutrition
MeSH Terms: interventions — Resistance Training; Diet, Ketogenic; Diet, Western

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ketogenic diet (Experimental): Participants will perform a single exercise bout after 4 weeks of resistance training combined with a ketogenic diet (KD group).
  Interventions: Other: resistance training; Other: ketogenic diet
- western diet (Active Comparator): Participants will perform a single exercise bout after 4 weeks of resistance training combined with a western diet (WD group).
  Interventions: Other: resistance training; Other: western diet

INTERVENTIONS:
Other: resistance training — All participants perform a four-day resistance training aimed to stimulate a hypertrophic response.
Other: ketogenic diet — Subjects allocated to the ketogenic diet arm (KD group) consume less than 50 g of carbohydrates per day.
  Arms: ketogenic diet
Other: western diet — Subjects allocated to the western diet arm (WD group) consume a standard diet based on 55% of their daily calories from carbohydrates.
  Arms: western diet

SUMMARY:
The purpose of this study is to investigate the effects of 4 weeks of carbohydrate deprivation (through a ketogenic diet) on hypertrophy signalling after a single bout of exercise in healthy trained male subjects, and the impact on body composition, muscle strength, and blood parameters.

ELIGIBILITY:
Inclusion Criteria:

* at least 2 years of resistance-training experience
* Body mass index: more than 18 kg/m2 and less than 30 kg/m2

Exclusion Criteria:

* metabolic diseases or noncommunicable diseases (cardiovascular, liver, respiratory, cancer, etc)
* experience with the ketogenic diet (last six months)
* acute inflammatory status
* treatment with steroids in the past 3 months

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-06-20 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
mammalian target of rapamycin (mTOR) signalling | Change from baseline to 4 weeks
  Measurement of the change in muscle protein anabolic signalling pathway in response to a single bout of resistance exercise by western blot analysis.

SECONDARY OUTCOMES:
Skeletal muscle mass | Change from baseline to 4 weeks
  Measurement of the change in kilograms of muscle mass via Dexa

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Paoli, MD, Principal Investigator — University of Padova
Locations (1):
- Nutex LAB, Padua, Italy

IPD SHARING:
Plan to Share IPD: No